CLINICAL TRIAL: NCT02764333
Title: A Phase II Trial of TPIV200/huFR-1 (A Multi-Epitope Anti-Folate Receptor Vaccine) Plus Anti-PD-L1 MEDI4736 (Durvalumab) in Patients With Platinum Resistant Ovarian Cancer
Brief Title: TPIV200/huFR-1 (A Multi-Epitope Anti-Folate Receptor Vaccine) Plus Anti-PD-L1 MEDI4736 (Durvalumab) in Patients With Platinum Resistant Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Marker Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-011
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-01

CONDITIONS: Ovarian Cancer
Keywords: TPIV200/huFR-1; Anti-PD-L1; vaccine; 16-011
MeSH Terms: conditions — Ovarian Neoplasms | interventions — durvalumab

ARMS (1):
- vaccine (Experimental): Patients will receive an intradermal (ID) injection of TPIV200 (500 μg per peptide) and GM-CSF (125 μg per peptide) on Day 1 of cycles 1-6. They will also receive intravenous (IV) injections of durvalumab (750mg) on Days 1 and 15 of cycles 1-12. Radiologic tumor assessment will be repeated every 12 weeks (or 3 cycles) during and after treatment, until time of progression. Treatment will continue until progression, intolerance, withdrawal, study completion, or study termination.
  Interventions: Biological: TPIV200; Biological: Durvalumab

INTERVENTIONS:
Biological: TPIV200
Biological: Durvalumab

SUMMARY:
This is a Phase 2 clinical trial, which tests two investigational drugs: TPIV200/huFR-1 (also called TPIV200), which is a vaccine consisting of proteins from the folate receptor alpha mixed with GM-CSF, and durvalumab (MEDI4736) , which is an antibody drug that help un-block parts of the immune system. The aim of this study is to find out whether these drugs, when given together are safe, and whether they are effective in treating cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have recurrent or persistent platinum-resistant epithelial ovarian, fallopian tube, or primary peritoneal carcinoma with measureable disease (as defined by RECIST 1.1.) who have received at least one prior platinum-based therapy.

Platinum-based therapy is defined as treatment with carboplatin, cisplatin or another organoplatinum compound.

Platinum-resistant is defined as having had disease progression within 6 months or most recent platinum therapy, or having disease progression while receiving previous platinum-based chemotherapy.

Histologic documentation of diagnosis of carcinoma is required and the following histologic subtypes are eligible: high grade serous, clear cell, endometrioid, carcinoma, adenocarcinoma, mixed (including above subtypes only).

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Resolution of (non-laboratory) adverse effects of recent surgery, radiotherapy, or chemotherapy to Grade ≤1 prior to first study treatment (with the exception of alopecia or neuropathy; chemotherapy-induced peripheral neuropathy up to Grade ≤2 will be permitted)
* Patients must have measurable disease. Measurable disease is defined by RECIST (version 1.1). Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and has not been previously irradiated. Each lesion must be ≥ 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or ≥ 20 mm when measured by chest x-ray. Lymph nodes must be ≥ 15 mm in short axis when measured by CT or MRI.
* Adequate normal organ and marrow function defined by the following laboratory results obtained within 14 days prior to first treatment:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (> 1500 per mm3)
  * Platelet ≥ 100 x 10^9/L (>100,000 per mm3)
  * Hemoglobin ≥ 9.0 g/dL
  * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). (Unless Gilbert's Syndrome, without concurrent clinically significant liver disease)
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
  * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Creatinine CL = Weight (kg) x (140 - Age) x 0.85 (mL/min) 72 x serum creatinine (mg/dL)

* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site); Previous enrollment in the present study.
* Participation in another clinical study with receipt of an investigational product during the last 4 weeks
* Any previous treatment with a PD-1 or PD-L1 inhibitor, including durvalumab
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease (eg, cervical cancer in situ)
  * Adequately treated stage 1 breast or stage 1 low grade endometrial cancer
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) < 21 days prior to the first dose of study drug.
* Mean QT interval corrected for heart rate (QTc) >/= 470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Steroid pre-medication for CT scan contrast or study drug, is allowable, regardless of dose.
* Any prior Grade >/= 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > Grade 1
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab or any excipient
* History of hypersensitivity to TPIV200
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
* Subjects who are pregnant, breast-feeding or of reproductive potential who are not employing an effective method of birth control
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Subjects with uncontrolled seizures
* Known hypersensitivity reaction to the GM-CSF adjuvant
* Patients who have developed any evidence of clinical or radiologic pneumonitis, COP/BOOP, or other lung injury, during treatment with prior FRα-targeting therapy, such as mirvetuximab soravtansine (IMGN853), or with any prior cancer immunotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Konner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center at Rockville, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine: Patients will receive an intradermal (ID) injection of TPIV200 (500 μg per peptide) and GM-CSF (125 μg per peptide) on Day 1 of cycles 1-6. They will also receive intravenous (IV) injections of durvalumab (750mg) on Days 1 and 15 of cycles 1-12. Radiologic tumor assessment will be repeated every 12 weeks (or 3 cycles) during and after treatment, until time of progression. Treatment will continue until progression, intolerance, withdrawal, study completion, or study termination.
  TPIV200
  Durvalumab
Period: Overall Study
Arm/Group | Vaccine
Started | 29
Completed | 28
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vaccine
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: (CR+PR) and will be assessed by RECIST 1.1. Pre-defined deviations from RECIST will be permitted to allow select patients deemed to be benefitting from treatment to receive continued therapy.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine
Number analyzed (Participants) | 29
Participants
  Partial Response | 1
  Stable Disease | 6
  Progression of Disease | 4
  Not Entered | 18

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Vaccine
All-Cause Mortality (participants affected / at risk) | 4/29
Serious Adverse Events (participants affected / at risk) | 9/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=29)
Breast pain (Reproductive system and breast disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Kidney infection (Infections and infestations) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Pain (General disorders) | 1
Platelet count decreased (Investigations) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=29)
Injection site reaction (General disorders) | 11
Nausea (Gastrointestinal disorders) | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Fatigue (General disorders) | 8
Constipation (Gastrointestinal disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Serum amylase increased (Investigations) | 3
Vomiting (Gastrointestinal disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bladder infection (Infections and infestations) | 2
Bloating (Gastrointestinal disorders) | 2
Hyperthyroidism (Endocrine disorders) | 2
Lipase increased (Investigations) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT02764333/Prot_SAP_000.pdf